CLINICAL TRIAL: NCT00242710
Title: A Double-Blind, Randomized, Placebo- And Active-Controlled Efficacy And Safety Study Of Bazedoxifene/Conjugated Estrogens Combinations For Prevention Of Endometrial Hyperplasia And Prevention Of Osteoporosis In Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene/Conjugated Estrogens Combinations In Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3115A1-304
Record Dates: First submitted 2005-10-18; First posted 2005-10-20 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-10

CONDITIONS: Endometrial Hyperplasia; Osteoporosis
Keywords: Endometrium; Uterus; Menopause
MeSH Terms: conditions — Endometrial Hyperplasia; Osteoporosis | interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): BZA 20mg/CE 0.625
  Interventions: Drug: Bazedoxifene/Conjugated Estrogen
- Arm 2 (Experimental): BZA 20mg/CE 0.45
  Interventions: Drug: Bazedoxifene/Conjugated Estrogen
- Arm 3 (Active Comparator): CE 0.45mg/MPA1.5mg
  Interventions: Drug: CE 0.45 mg/MPA 1.5mg
- Arm 4 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bazedoxifene/Conjugated Estrogen — Subjects will take 1 capsule orally, once daily, at approximately the same time each day continuously for the duration of the study.
  Arms: 1
Drug: Bazedoxifene/Conjugated Estrogen — Subjects will take 1 capsule orally, once daily, at approximately the same time each day continuously for the duration of the study.
  Arms: Arm 2
Drug: CE 0.45 mg/MPA 1.5mg — Subjects will take 1 capsule orally, once daily, at approximately the same time each day continuously for the duration of the study.
  Arms: Arm 3
Other: Placebo — Subjects will take 1 capsule orally, once daily, at approximately the same time each day continuously for the duration of the study.
  Arms: Arm 4

SUMMARY:
The purpose of this study is to determine whether bazedoxifene/conjugated estrogens combinations are effective for the prevention of endometrial hyperplasia and for the prevention of osteoporosis in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women, aged 40 to less than 65 years
* Intact uterus
* At least 12 months of spontaneous amenorrhea, OR 6 months spontaneous amenorrhea with follicle-stimulating hormone (FSH) levels > 40 mIU/mL.

Exclusion Criteria:

* Use of oral estrogen-, progestin-, androgen-, or SERM-containing drug products within 8 weeks before screening (12 weeks for the osteoporosis substudy)
* A history or active presence of clinically important medical disease
* Malabsorption disorders

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1083 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Inverness, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3115A1-304&StudyName=Study%20Evaluating%20Bazedoxifene/Conjugated%20Estrogens%20Combinations%20In%20Postmenopausal%20Women

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This main study also included osteoporosis substudy only for the purpose of the assessment of relevant parameters.
Groups:
- Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg: Bazedoxifene 20 milligram (mg)/conjugated estrogen 0.45 mg capsule orally once daily at approximately the same time each day continuously up to Year 1 during the core study and up to Year 2 during the study extension. Participants also received Caltrate plus D tablet containing calcium 600 mg and vitamin D 200 international unit (IU) orally once daily up to Year 2.
- Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg: Bazedoxifene 20 mg/conjugated estrogen 0.625 mg capsule orally once daily at approximately the same time each day continuously up to Year 1 during the core study and up to Year 2 during the study extension. Participants also received Caltrate plus D tablet containing calcium 600 mg and vitamin D 200 IU orally once daily up to Year 2.
- Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg: Conjugated estrogen 0.45 mg/medroxyprogesterone acetate 1.5 mg capsule orally once daily at approximately the same time each day continuously up to Year 1 during the core study and up to Year 2 during the study extension. Participants also received Caltrate plus D tablet containing calcium 600 mg and vitamin D 200 IU orally once daily up to Year 2.
- Placebo: Placebo matched to bazedoxifene/conjugated estrogen or conjugated estrogen/medroxyprogesterone acetate capsule orally once daily at approximately the same time each day continuously up to Year 1 during the core study and up to Year 2 during the study extension. Participants also received Caltrate plus D tablet containing calcium 600 mg and vitamin D 200 IU orally once daily up to Year 2.
Period: Core Study (up to Year 1)
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Started | 373 | 353 | 183 | 174
Treated | 361 | 349 | 179 | 172
Completed | 287 | 289 | 132 | 143
Not Completed | 86 | 64 | 51 | 31
Not completed — Adverse Event | 30 | 25 | 23 | 14
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 8 | 8 | 7 | 3
Not completed — Other | 6 | 1 | 0 | 2
Not completed — Protocol Violation | 2 | 9 | 1 | 3
Not completed — Withdrawal by Subject | 27 | 16 | 15 | 6
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Randomized but not Treated | 12 | 4 | 4 | 2
Period: Period Between Core Study and Extension
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Started | 287 | 289 | 132 | 143
Completed | 168 | 177 | 84 | 94
Not Completed | 119 | 112 | 48 | 49
Not completed — Adverse Event | 2 | 3 | 5 | 2
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Other | 24 | 24 | 9 | 11
Not completed — Extension not Available | 17 | 21 | 8 | 7
Not completed — Protocol Violation | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 75 | 63 | 24 | 28
Period: Study Extension (up to Year 2)
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Started | 168 | 177 | 84 | 94
Completed | 141 | 148 | 69 | 84
Not Completed | 27 | 29 | 15 | 10
Not completed — Adverse Event | 7 | 9 | 2 | 4
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 7 | 7 | 5 | 0
Not completed — Other | 3 | 5 | 4 | 3
Not completed — Protocol Violation | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 6 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomly assigned participants who took at least 1 dose of test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo | Total
Number analyzed (Participants) | 361 | 349 | 179 | 172 | 1061
Age Continuous [Mean (Standard Deviation); unit: years] | 54.62 (4.74) | 54.44 (4.62) | 54.30 (4.56) | 54.19 (4.62) | 54.44 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 361 | 349 | 179 | 172 | 1061
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hyperplasia at Screening
Description: Endometrial hyperplasia was assessed by endometrial biopsies. All endometrial biopsies were read centrally by 2 primary pathologists. Participants were considered to have a diagnosis of hyperplasia if both pathologists read hyperplasia (simple hyperplasia with or without atypia or complex hyperplasia with or without atypia). If the both pathologists disagreed on the presence of hyperplasia, a third pathologist was consulted, with the final diagnosis determined by the majority opinion.
Time Frame: Screening
Population: Endometrial hyperplasia at screening was an exclusion criterion and participants who had hyperplasia were not included in the analysis. Therefore this data is not available.
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Hyperplasia at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: Efficacy evaluable (EE) analysis population for Year 1: all participants who were randomized and took at least 1 dose of test article, who had a screening endometrial biopsy with readings by at least 2 blinded central pathologists, had a biopsy during Month 12, or had hyperplasia diagnosed before Month 12 and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 261 | 273 | 119 | 135
percentage of participants | 0.00 [0.00 to 1.14] | 1.10 [0.30 to 2.82] | 0.00 [0.00 to 2.49] | 0.00 [0.00 to 2.19]

3. Primary Outcome: Bone Mineral Density (BMD) of Lumbar Spine at Screening
Description: BMD measurements of the anteroposterior lumbar spine were acquired by dual-energy x-ray absorptiometry (DXA), twice during screening in participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. An average of the 2 readings was reported.
Time Frame: Screening
Population: Modified intent-to-treat (MITT) population for BMD of lumber spine included all randomized participants took at least 1 dose of test article, and had a baseline and at least 1 on-therapy evaluation of BMD (scans acquired more than 60 days after the test article administration was stopped were excluded) at Year 1.
Measure: Mean (Standard Deviation); unit: grams per square centimeter (g/cm^2)
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 146 | 144 | 60 | 65
grams per square centimeter (g/cm^2) | 1.00 (0.12) | 1.01 (0.12) | 1.02 (0.12) | 1.01 (0.12)

4. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Lumbar Spine at Month 12
Description: BMD measurements of the anteroposterior lumbar spine were acquired by DXA, twice at Month 12 in participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. An average of the 2 readings was reported.
Time Frame: Baseline, Month 12
Population: MITT population for BMD of lumber spine: all randomized participants who took at least 1 dose of test article, and had a baseline and at least 1 on-therapy evaluation of BMD (scans acquired more than 60 days after test article administration was stopped were excluded) at Year 1. Missing values imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 146 | 144 | 60 | 65
percent change | 0.80 (0.24) | 0.80 (0.24) | 2.22 (0.37) | -1.56 (0.35)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; An analysis of covariance (ANCOVA) model was used with treatment and center as main effects and baseline BMD and years since menopause as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; Least Squares (LS) Mean Difference = 2.37, 95% CI 2-sided [1.56 to 3.18]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; An ANCOVA model was used with treatment and center as main effects and baseline BMD and years since menopause as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.36, 95% CI 2-sided [1.56 to 3.17]
Statistical Analysis 3: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.78, 95% CI 2-sided [2.81 to 4.76]

5. Primary Outcome: Bone Mineral Density (BMD) of Total Hip at Screening
Description: BMD measurements of the total hip were acquired by DXA, twice during screening in participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. An average of the 2 readings was reported.
Time Frame: Screening
Population: MITT population for BMD of total hip included all randomized participants who took at least 1 dose of test article, and had a baseline and at least 1 on-therapy evaluation of BMD (scans acquired more than 60 days after the test article administration was stopped were excluded) at Year 1. Missing values were imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 148 | 145 | 60 | 66
g/cm^2 | 0.90 (0.11) | 0.89 (0.11) | 0.90 (0.10) | 0.89 (0.11)

6. Primary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Total Hip at Month 12
Description: BMD measurements of the total hip were acquired by DXA, twice at Month 12 in participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. An average of the 2 readings was reported.
Time Frame: Baseline, Month 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 148 | 145 | 60 | 66
percent change | 0.62 (0.19) | 0.84 (0.19) | 1.47 (0.29) | -0.99 (0.27)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.61, 95% CI 2-sided [0.97 to 2.24]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.82, 95% CI 2-sided [1.19 to 2.46]
Statistical Analysis 3: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.46, 95% CI 2-sided [1.69 to 3.23]

7. Secondary Outcome: Percentage of Days With Breast Pain
Description: Percentage of days with breast pain in each 4-week period (for example, Week 1 to 4, 5 to 8) calculated as the number of days on which a participants reported breast pain divided by total number of days with data recorded multiplied by 100. Data was collected every day after randomization up to Year 1 and was analyzed in 4 weeks intervals. Data for screening was not analyzed since data were collected only for 7 days at screening which was not considered comparable to 4-week post-baseline data.
Time Frame: Screening, Week 1 to 4, 5 to 8, 9 to 12, 13 to 16, 17 to 20, 21 to 24, 25 to 28, 29 to 32, 33 to 36, 37 to 40, 41 to 44, 45 to 48, 49 to 52
Population: MITT population for breast pain: all randomized participants who took at least 1 dose of test article, and had data available at least for 5 of 7 days at screening and 20 days for at least 1 post-baseline interval. n=participants evaluable at specified time periods for each arm, respectively.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 347 | 329 | 168 | 163
percentage of days
  Week 1-4 (n=347, 329, 168, 163) | 1.55 (0.49) | 1.22 (0.51) | 3.49 (0.65) | 0.89 (0.66)
  Week 5-8 (n=331, 323, 158, 158) | 1.71 (0.68) | 1.58 (0.68) | 5.54 (0.91) | 1.36 (0.92)
  Week 9-12 (n=323, 317, 150, 152) | 2.00 (0.68) | 1.01 (0.68) | 4.80 (0.93) | 1.36 (0.92)
  Week 13-16 (n=315, 310, 141, 150) | 1.87 (0.60) | 0.88 (0.61) | 3.92 (0.84) | 0.77 (0.81)
  Week 17-20 (n=313, 309, 141, 149) | 2.11 (0.63) | 1.57 (0.64) | 4.23 (0.88) | 1.61 (0.85)
  Week 21-24 (n=312, 306, 141, 147) | 2.49 (0.78) | 1.85 (0.79) | 5.01 (1.08) | 1.26 (1.06)
  Week 25-28 (n=306, 298, 136, 144) | 2.60 (0.77) | 1.31 (0.78) | 4.91 (1.07) | 1.39 (1.04)
  Week 29-32 (n=301, 297, 133, 143) | 1.80 (0.62) | 0.82 (0.63) | 3.98 (0.87) | 0.17 (0.84)
  Week 33-36 (n=297, 294, 132, 143) | 1.29 (0.57) | 0.25 (0.58) | 3.49 (0.80) | -0.26 (0.77)
  Week 37-40 (n=295, 288, 130, 140) | 1.61 (0.62) | 0.25 (0.64) | 3.87 (0.88) | 0.57 (0.85)
  Week 41-44 (n=286, 285, 128, 140) | 1.99 (0.66) | 0.56 (0.67) | 2.49 (0.92) | 0.86 (0.89)
  Week 45-48 (n=282, 284, 127, 140) | 1.68 (0.67) | 1.26 (0.68) | 2.52 (0.94) | 1.17 (0.90)
  Week 49-52 (n=170, 171, 70, 91) | 1.07 (1.12) | 1.68 (1.16) | 5.27 (1.69) | 1.49 (1.50)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 1-4: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.373, ANCOVA; LS Mean Difference = 0.66, 95% CI 2-sided [-0.80 to 2.12]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 5-8: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.738, ANCOVA; LS Mean Difference = 0.35, 95% CI 2-sided [-1.70 to 2.40]
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 9-12: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.539, ANCOVA; LS Mean Difference = 0.65, 95% CI 2-sided [-1.41 to 2.71]
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 13-16: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.233, ANCOVA; LS Mean Difference = 1.09, 95% CI 2-sided [-0.71 to 2.90]
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 17-20: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.605, ANCOVA; LS Mean Difference = 0.50, 95% CI 2-sided [-1.39 to 2.39]
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 21-24: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.305, ANCOVA; LS Mean Difference = 1.23, 95% CI 2-sided [-1.12 to 3.57]
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 25-28: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.299, ANCOVA; LS Mean Difference = 1.22, 95% CI 2-sided [-1.08 to 3.52]
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 29-32: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.092, ANCOVA; LS Mean Difference = 1.62, 95% CI 2-sided [-0.27 to 3.51]
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 33-36: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.080, ANCOVA; LS Mean Difference = 1.55, 95% CI 2-sided [-0.18 to 3.29]
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 37-40: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.279, ANCOVA; LS Mean Difference = 1.04, 95% CI 2-sided [-0.85 to 2.92]
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 41-44: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.260, ANCOVA; LS Mean Difference = 1.13, 95% CI 2-sided [-0.84 to 3.11]
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 45-48: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.618, ANCOVA; LS Mean Difference = 0.51, 95% CI 2-sided [-1.50 to 2.52]
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 49-52: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.810, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-3.78 to 2.96]
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 1-4: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.654, ANCOVA; LS Mean Difference = 0.34, 95% CI 2-sided [-1.14 to 1.81]
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 5-8: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.834, ANCOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-1.84 to 2.28]
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 9-12: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.744, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-2.41 to 1.72]
Statistical Analysis 17: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 13-16: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.909, ANCOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-1.70 to 1.91]
Statistical Analysis 18: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 17-20: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.963, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-1.94 to 1.85]
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 21-24: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.625, ANCOVA; LS Mean Difference = 0.59, 95% CI 2-sided [-1.77 to 2.94]
Statistical Analysis 20: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 25-28: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.947, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-2.39 to 2.23]
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 29-32: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.505, ANCOVA; LS Mean Difference = 0.64, 95% CI 2-sided [-1.25 to 2.53]
Statistical Analysis 22: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 33-36: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.564, ANCOVA; LS Mean Difference = 0.51, 95% CI 2-sided [-1.23 to 2.25]
Statistical Analysis 23: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 37-40: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.739, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-2.21 to 1.57]
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 41-44: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.766, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-2.27 to 1.67]
Statistical Analysis 25: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 45-48: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.931, ANCOVA; LS Mean Difference = 0.09, 95% CI 2-sided [-1.92 to 2.10]
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 49-52: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.911, ANCOVA; LS Mean Difference = 0.19, 95% CI 2-sided [-3.17 to 3.56]
Statistical Analysis 27: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 1-4: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.003, ANCOVA; LS Mean Difference = 2.61, 95% CI 2-sided [0.92 to 4.30]
Statistical Analysis 28: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 5-8: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.18, 95% CI 2-sided [1.79 to 6.58]
Statistical Analysis 29: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 9-12: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.005, ANCOVA; LS Mean Difference = 3.45, 95% CI 2-sided [1.03 to 5.86]
Statistical Analysis 30: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 13-16: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = 3.15, 95% CI 2-sided [1.01 to 5.30]
Statistical Analysis 31: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 17-20: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.023, ANCOVA; LS Mean Difference = 2.61, 95% CI 2-sided [0.36 to 4.87]
Statistical Analysis 32: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 21-24: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.008, ANCOVA; LS Mean Difference = 3.75, 95% CI 2-sided [0.96 to 6.54]
Statistical Analysis 33: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 25-28: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.012, ANCOVA; LS Mean Difference = 3.52, 95% CI 2-sided [0.78 to 6.26]
Statistical Analysis 34: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 29-32: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.81, 95% CI 2-sided [1.55 to 6.07]
Statistical Analysis 35: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 33-36: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.75, 95% CI 2-sided [1.68 to 5.83]
Statistical Analysis 36: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 37-40: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.004, ANCOVA; LS Mean Difference = 3.30, 95% CI 2-sided [1.05 to 5.54]
Statistical Analysis 37: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 41-44: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.175, ANCOVA; LS Mean Difference = 1.63, 95% CI 2-sided [-0.73 to 3.99]
Statistical Analysis 38: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 45-48: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.270, ANCOVA; LS Mean Difference = 1.35, 95% CI 2-sided [-1.05 to 3.75]
Statistical Analysis 39: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 49-52: An ANCOVA model was used with treatment, center as factors, and baseline as the covariate; Test type: Superiority or Other; p = 0.077, ANCOVA; LS Mean Difference = 3.78, 95% CI 2-sided [-0.41 to 7.97]

8. Secondary Outcome: Percentage of Participants With Uterine Bleeding or Spotting
Description: Data was collected every day after randomization up to Year 1 and was analyzed in 4 weeks intervals. Data for screening was not analyzed since data were collected only for 7 days at screening which was not considered comparable to 4-week post-baseline data.
Time Frame: as for outcome 7
Population: MITT population for uterine bleeding or spotting included all randomized participants who had received at least 1 dose of test article and had at least 1 day of on-therapy bleeding data. Imputation=LOCF. n=participants evaluable for this measure at specified time periods for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 330 | 315 | 159 | 155
percentage of participants
  Week 1-4 (n=330, 313, 159, 155) | 5.45 | 4.15 | 19.50 | 4.52
  Week 5-8 (n=320, 315, 153, 151) | 2.19 | 2.86 | 23.53 | 3.31
  Week 9-12 (n=316, 310, 147, 146) | 2.53 | 4.52 | 25.17 | 2.74
  Week 13-16 (n=310, 296, 137, 149) | 2.90 | 2.70 | 16.79 | 1.34
  Week 17-20 (n=315, 311, 144, 150) | 2.22 | 1.61 | 16.67 | 0.67
  Week 21-24 (n=311, 306, 142, 147) | 0.96 | 1.31 | 16.20 | 2.72
  Week 25-28 (n=294, 290, 131, 143) | 2.04 | 1.38 | 9.92 | 2.10
  Week 29-32 (n=298, 297, 135, 141) | 0.67 | 2.02 | 11.11 | 0.71
  Week 33-36 (n=296, 291, 134, 140) | 2.03 | 2.75 | 11.94 | 2.86
  Week 37-40 (n=282, 279, 131, 139) | 2.13 | 2.87 | 11.45 | 2.88
  Week 41-44 (n=285, 284, 132, 141) | 1.40 | 1.06 | 8.33 | 2.84
  Week 45-48 (n=280, 282, 130, 140) | 1.79 | 2.48 | 11.54 | 2.86
  Week 49-52 (n=45, 51, 15, 31) | 0.00 | 1.96 | 33.33 | 6.45
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.826, Fisher Exact
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.534, Fisher Exact
Statistical Analysis 3: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 4: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.516, Fisher Exact
Statistical Analysis 5: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.446, Fisher Exact
Statistical Analysis 6: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.218, Fisher Exact
Statistical Analysis 7: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 8: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 9: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.733, Fisher Exact
Statistical Analysis 10: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.736, Fisher Exact
Statistical Analysis 11: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.449, Fisher Exact
Statistical Analysis 12: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.489, Fisher Exact
Statistical Analysis 13: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.163, Fisher Exact
Statistical Analysis 14: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.813, Fisher Exact
Statistical Analysis 15: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.777, Fisher Exact
Statistical Analysis 16: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.448, Fisher Exact
Statistical Analysis 17: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.507, Fisher Exact
Statistical Analysis 18: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.669, Fisher Exact
Statistical Analysis 19: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.281, Fisher Exact
Statistical Analysis 20: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.689, Fisher Exact
Statistical Analysis 21: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.437, Fisher Exact
Statistical Analysis 22: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 23: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 24: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.227, Fisher Exact
Statistical Analysis 25: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.758, Fisher Exact
Statistical Analysis 26: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.554, Fisher Exact
Statistical Analysis 27: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 1-4: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 28: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 5-8: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 29: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 9-12: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 30: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 13-16: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 31: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 17-20: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 32: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 21-24: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 33: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 25-28: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.008, Fisher Exact
Statistical Analysis 34: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 29-32: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 35: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 33-36: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.005, Fisher Exact
Statistical Analysis 36: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 37-40: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.008, Fisher Exact
Statistical Analysis 37: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 41-44: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.062, Fisher Exact
Statistical Analysis 38: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 45-48: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.007, Fisher Exact
Statistical Analysis 39: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; Week 49-52: The Fisher exact test was used for comparisons between groups; Test type: Superiority or Other; p = 0.029, Fisher Exact

9. Secondary Outcome: Percentage of Participants With Hyperplasia at Month 24
Description: as for outcome 1
Time Frame: Month 24
Population: EE analysis population for Year 2 included all randomized participants who took at least 1 dose of test article, participated in study extension, had a screening endometrial biopsy with readings by at least 2 blinded central pathologists, had biopsy during Month 24, or had hyperplasia diagnosed before Month 24 and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 131 | 142 | 66 | 79
percentage of participants | 0.00 [0.00 to 2.78] | 4.93 [2.00 to 9.89] | 0.00 [0.00 to 5.44] | 0.00 [0.00 to 4.56]

10. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Lumbar Spine at Month 24
Description: BMD measurements of the anteroposterior lumbar spine were acquired by DXA, twice at Month 24 in participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. An average of the 2 readings was reported.
Time Frame: Baseline, Month 24
Population: MITT population for BMD of lumber spine: all participants who took at least 1 dose of test article, participated in study extension, and had a baseline and at least 1 on-therapy evaluation of BMD (scans acquired more than 60 days after the test article administration was stopped were excluded) at Year 2. Missing values imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 87 | 87 | 40 | 39
percent change | 0.96 (0.40) | 0.86 (0.41) | 2.39 (0.57) | -2.29 (0.57)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.25, 95% CI 2-sided [1.92 to 4.58]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 3.14, 95% CI 2-sided [1.83 to 4.46]
Statistical Analysis 3: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 4.68, 95% CI 2-sided [3.13 to 6.23]

11. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of Total Hip at Month 24
Description: BMD measurements of the total hip were acquired by DXA, twice at Month 24 in participants who entered the osteoporosis substudy. The second scan was to be performed on the same day as the first; however, the participant was to be removed completely from the table after the first scan and repositioned for the second scan. An average of the 2 readings was reported.
Time Frame: Baseline, Month 24
Population: MITT population for BMD of total hip: all participants who took at least 1 dose of test article, participated in study extension, and had a baseline and at least 1 on-therapy evaluation of BMD (scans acquired more than 60 days after the test article administration was stopped were excluded) at Year 2. Missing values imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Number analyzed (Participants) | 87 | 88 | 40 | 39
percent change | 0.30 (0.31) | 0.41 (0.32) | 0.85 (0.44) | -1.53 (0.45)
Statistical Analysis 1: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.83, 95% CI 2-sided [0.80 to 2.87]
Statistical Analysis 2: Comparison: Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 1.94, 95% CI 2-sided [0.92 to 2.97]
Statistical Analysis 3: Comparison: Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; LS Mean Difference = 2.38, 95% CI 2-sided [1.17 to 3.59]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg | Placebo
Serious Adverse Events (participants affected / at risk) | 22/361 | 19/349 | 7/179 | 7/172
Other Adverse Events (participants affected / at risk) | 322/361 | 309/349 | 165/179 | 152/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg (N=361) | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg (N=349) | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg (N=179) | Placebo (N=172)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Biopsy endometrium abnormal (Investigations) | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 0
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bazedoxifene 20 mg/Conjugated Estrogen 0.45 mg (N=361) | Bazedoxifene 20 mg/Conjugated Estrogen 0.625 mg (N=349) | Conjugated Estrogen 0.45 mg/Medroxyprogesterone Acetate 1.5mg (N=179) | Placebo (N=172)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 5 | 2 | 4
Palpitations (Cardiac disorders) | 7 | 0 | 2 | 4
Ear pain (Ear and labyrinth disorders) | 3 | 4 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 7 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 5 | 6 | 8 | 3
Abdominal pain (Gastrointestinal disorders) | 20 | 28 | 17 | 5
Abdominal pain lower (Gastrointestinal disorders) | 10 | 17 | 9 | 3
Abdominal pain upper (Gastrointestinal disorders) | 32 | 22 | 12 | 7
Constipation (Gastrointestinal disorders) | 23 | 16 | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 21 | 22 | 11 | 14
Dyspepsia (Gastrointestinal disorders) | 19 | 21 | 11 | 18
Flatulence (Gastrointestinal disorders) | 2 | 7 | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 7 | 2 | 2
Nausea (Gastrointestinal disorders) | 25 | 20 | 14 | 10
Stomach discomfort (Gastrointestinal disorders) | 8 | 10 | 7 | 4
Toothache (Gastrointestinal disorders) | 19 | 19 | 12 | 4
Vomiting (Gastrointestinal disorders) | 11 | 10 | 8 | 5
Fatigue (General disorders) | 10 | 13 | 7 | 8
Non-cardiac chest pain (General disorders) | 6 | 7 | 4 | 7
Oedema peripheral (General disorders) | 9 | 10 | 4 | 4
Pain (General disorders) | 17 | 15 | 3 | 12
Pyrexia (General disorders) | 4 | 5 | 4 | 6
Hypersensitivity (Immune system disorders) | 10 | 9 | 3 | 2
Seasonal allergy (Immune system disorders) | 11 | 7 | 5 | 5
Bronchitis (Infections and infestations) | 17 | 18 | 7 | 13
Gastroenteritis (Infections and infestations) | 6 | 10 | 9 | 4
Gastroenteritis viral (Infections and infestations) | 11 | 12 | 6 | 3
Influenza (Infections and infestations) | 43 | 35 | 24 | 14
Localised infection (Infections and infestations) | 2 | 4 | 4 | 1
Nasopharyngitis (Infections and infestations) | 83 | 82 | 42 | 30
Onychomycosis (Infections and infestations) | 2 | 4 | 5 | 1
Oral herpes (Infections and infestations) | 3 | 4 | 5 | 1
Pharyngitis (Infections and infestations) | 11 | 7 | 6 | 6
Sinusitis (Infections and infestations) | 32 | 23 | 9 | 13
Tooth abscess (Infections and infestations) | 7 | 7 | 4 | 7
Tooth infection (Infections and infestations) | 5 | 7 | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 29 | 35 | 15 | 12
Urinary tract infection (Infections and infestations) | 26 | 21 | 11 | 9
Vulvovaginal mycotic infection (Infections and infestations) | 12 | 20 | 16 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 6 | 8 | 3 | 1
Back injury (Injury, poisoning and procedural complications) | 4 | 7 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 8 | 3 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 1 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 7 | 2 | 2
Joint sprain (Injury, poisoning and procedural complications) | 8 | 8 | 3 | 2
Muscle strain (Injury, poisoning and procedural complications) | 4 | 6 | 3 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 8 | 5 | 4 | 2
Procedural pain (Injury, poisoning and procedural complications) | 16 | 20 | 9 | 12
Weight increased (Investigations) | 10 | 8 | 4 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 3 | 5 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 14 | 6 | 6 | 13
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 56 | 22 | 28
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 9 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 60 | 66 | 33 | 23
Muscle spasms (Musculoskeletal and connective tissue disorders) | 37 | 29 | 16 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 13 | 8 | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7 | 7 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 34 | 28 | 16 | 16
Neck pain (Musculoskeletal and connective tissue disorders) | 17 | 17 | 11 | 14
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 1 | 2 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 39 | 39 | 19 | 27
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4 | 1
Dizziness (Nervous system disorders) | 13 | 19 | 11 | 5
Headache (Nervous system disorders) | 94 | 78 | 58 | 41
Migraine (Nervous system disorders) | 7 | 11 | 6 | 3
Sciatica (Nervous system disorders) | 3 | 3 | 0 | 4
Sinus headache (Nervous system disorders) | 28 | 14 | 5 | 9
Tension headache (Nervous system disorders) | 1 | 2 | 4 | 3
Anxiety (Psychiatric disorders) | 10 | 4 | 7 | 6
Depression (Psychiatric disorders) | 6 | 9 | 6 | 7
Insomnia (Psychiatric disorders) | 25 | 17 | 10 | 13
Haematuria (Renal and urinary disorders) | 2 | 3 | 3 | 5
Breast pain (Reproductive system and breast disorders) | 18 | 18 | 19 | 7
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 7 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 5 | 7 | 4 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 18 | 29 | 28 | 10
Metrorrhagia (Reproductive system and breast disorders) | 9 | 4 | 10 | 4
Uterine haemorrhage (Reproductive system and breast disorders) | 2 | 2 | 7 | 1
Uterine spasm (Reproductive system and breast disorders) | 4 | 2 | 7 | 1
Vaginal discharge (Reproductive system and breast disorders) | 7 | 10 | 6 | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 13 | 18 | 22 | 4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 7 | 5 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 20 | 17 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 6 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 19 | 11 | 16
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 6 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 | 7 | 5 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 7 | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 16 | 7 | 6
Hot flush (Vascular disorders) | 38 | 37 | 11 | 7
Hypertension (Vascular disorders) | 14 | 11 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.